CLINICAL TRIAL: NCT05866120
Title: Effects of Physical Therapy on Land and Aquatic Physical Therapy on the Motor Function of Individuals With Parkinson's Disease
Brief Title: Effects of Land and Water Physiotherapy on Motor Function in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Clinical Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Função_Motora_DP+FA+FS
Record Dates: First submitted 2023-04-15; First posted 2023-05-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Physical Therapy Modalities; Muscle Strength; Aquatic Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals with Parkinson's Disease to perform physiotherapy on the ground. (Active Comparator): The protocols will last for 12 weeks, with a frequency of 2 times a week.
  Interventions: Other: Aquatic physiotherapy
- Individuals with Parkinson's Disease to undergo aquatic physiotherapy (Active Comparator): The protocols will last for 12 weeks, with a frequency of 2 times a week.
  Interventions: Other: Physiotherapy on the ground

INTERVENTIONS:
Other: Physiotherapy on the ground — Physical therapy will be performed on the ground, in 12 weeks, twice a week. The exercises will be based on a protocol developed by the researchers. This protocol has 15 exercises, aimed at muscle function and extensor musculature. All exercises can be adapted according to the severity of the individual, as well as the progression of these exercises will be made according to the adaptation and ease of individuals throughout the intervention.
  Arms: Individuals with Parkinson's Disease to undergo aquatic physiotherapy
Other: Aquatic physiotherapy — Aquatic physiotherapy will be performed in 12 weeks, twice a week, in shallow water. The exercises will be based on a protocol developed by the researchers. This protocol has 15 exercises, aimed at muscle function and extensor musculature. All exercises can be adapted according to the severity of the individual, as well as the progression of these exercises will be made according to the adaptation and ease of individuals throughout the intervention.
  Arms: Individuals with Parkinson's Disease to perform physiotherapy on the ground.

SUMMARY:
The aim of this study is to assess the effect of dry soil therapy and shallow water therapy on motor function in individuals with Parkinson's disease. Regarding the benefits, is there a difference between the therapies?

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic progressive neurological disorder that involves motor and non-motor symptoms that commonly include bradykinesia, rigidity, tremor and postural instability and culminates in functional decline and disability. Postural instability is due to postural alterations that are commonly found in these individuals. Muscular disorders characterized by the inability to generate adequate synergy patterns may be responsible for postural instability, leading to postural alterations in the sagittal plane, often with the onset of hyperkyphosis. Exercise is increasingly being recognized as an effective and highly promising non-pharmacological intervention to improve muscle strength in PD. Typical land-based physical therapy treatment includes strength training, gait and balance training and has several benefits in reducing motor symptoms of PD. Interventions such as aquatic physical therapy have a growing body of evidence to support the efficacy of exercise in the PD population. Aquatic exercise has the intrinsic advantage of helping individuals lose body weight, leading to greater efficacy of the exercise itself. Knowing that muscle strength is associated with functional capacity and disease severity, physiotherapy becomes an important treatment resource with exercises to improve muscle strength and consequently reduce subsequent functional difficulties. However, due to the scattered evidence of physiotherapy in PD, there is insufficient evidence to prescribe a defined rehabilitation program for strengthening the trunk extensor muscles. Although there is increasing evidence of the effectiveness of land-based or aquatic therapies, the evidence is insufficient to support or refute the effectiveness of one physiotherapy intervention over another. Therefore, this study aims to describe and compare the effects of 12 weeks of land-based physical therapy and aquatic physical therapy on the motor function of individuals with PD, as well as to evaluate muscle strength, functional capacity, mobility, flexibility, muscle mass and balance, while examining the linear relationship between PD severity and these parameters. A Randomized Clinical Trial will be conducted, which will include individuals diagnosed with Parkinson's Disease, akinetic-rigid type, with postural instability, classified from 1 to 3 on the Hoehn and Yahr Scale, aged between 50 and 85 years, who sign the Free and Informed Consent Form, and have a minimum score of 26 on the Montreal Cognitive Assessment (MoCA).

Individuals will be randomized into two treatment groups: land-based physiotherapy and aquatic physiotherapy. The evaluation will be carried out in two stages: pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's Disease and rated from 1 to 3 on the Hoehn and Yahr Scale;
* With akinetic rigid type PD;
* Aged between 50 and 85 years old;
* Minimum score of 26 on the Montreal Cognitive Assessment (MoCA);
* Who sign the Free and Informed Consent Term (TCLE).

Exclusion Criteria:

* Parkinson's disease of the dominant tremor type;
* Previous associated neurological diseases;
* Severe heart diseases;
* Uncontrolled high blood pressure;
* Previous spine surgeries;
* Inflammatory diseases of the spine;
* Chlorine allergy;
* Aquaphobia.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
MDS UPDRS Motor Assessment | 3 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a tool used to monitor the progression of the disease. Part II of the scale is the patient's self-assessment of daily activities, while part III is the motor assessment monitored by the clinician.
  Part II of the UPDRS assesses: speech, swallowing, writing, dressing, hygiene, falls, salivation, turning over in bed, walking, and cutting food.
  Part III of the UPDRS is the motor assessment monitored by clinical aspects and the cutoff points for classifying motor impairment as mild, moderate, and severe are as follows: Mild/Moderate - 32/33, Moderate/Severe - 58/59.
Berg Scale and Romberg Test | 3 months
  The Berg Balance Scale (BBS), translated and validated into Brazilian Portuguese in 2004, will be used to assess postural balance. The BBS, developed in 1992, consists of 14 common tasks involving static and dynamic balance. The tasks are evaluated through observation, presenting an ordinal scale of five alternatives, ranging from zero to four, totaling a maximum score of 56 points. The score decreases if the time to perform the task is not reached, or the individual needs supervision or external support to perform it.
  The Romberg test, on the other hand, consists of a clinical evaluation that reveals alterations in the patient's static balance, allowing the analysis of 3 neurophysiological bases that make balance possible: vestibular, visual and proprioceptive systems. This test exists to investigate disturbances that interfere with this task. A positive Romberg can be seen with loss of balance during the procedure.
Timed Up and Go (TUG) | 3 months
  The Timed Up and Go (TUG) test will also be used, which was developed to assess balance, risk of falls and functional capacity of elderly individuals, timing the time it takes the individual to leave the sitting position with the back supported on a chair, stand up, walk 3 meters to a marked point on the ground as fast as possible, turn around, return to the chair and sit down again, leaning against it. Performance is evaluated according to the time taken to perform the task. It takes approximately 1 to 2 minutes and only requires a chair approximately 46cm high and 65cm high armrest, a stopwatch and a 3 meter runner. The patient will perform the test a first time to understand the task and a second time for registration and evaluation. A time greater than 30 seconds to perform the task is indicative of the individual's functional dependence.
Dual-energy X-ray absorptiometry | 3 months
  Whole-body dual-energy X-ray absorptiometry (DEXA) is a sensitive and accurate method for quantifying body composition, including fat mass and lean body mass as a surrogate measure of skeletal muscle. Body composition will be estimated by dual-energy X-ray absorptiometry. Prior to scanning, participants will be asked to remove all removable objects containing metal (i.e. jewelry, glasses, clothing with buttons and/or zippers). Scans will be performed with participants lying supine along the longitudinal axis of the centerline of the scanning table. The feet will be tied together to immobilize the legs, while the hands will be kept in a prone position within the scanning region. All exams will be performed by the same evaluator. DEXA results will include body composition parameters including fat free mass, body fat percentage, fat mass and bone mineral density (whole body, whole left femur and lumbar spine vertebrae).
Ultrasonography | 3 months
  Ultrasonography is a non-invasive method for assessing the thickness and echogenicity of skeletal muscle. The research subjects will be approved to evaluate the quadriceps femoris musculature through Ultrasonography Nemio XG (Toshiba, Japan) in B mode and a 3.75 MHz convex transducer.
  The transducer will be coated with a water-soluble transmission gel to provide acoustic contact without depressing the dermal surface.
Isokinetic dynamometer - torque | 3 months
  The isokinetic dynamometer is considered the gold standard instrument for assessing muscle performance, whether to analyze the effectiveness of training, treatment or even to verify a person's muscle condition. The individuals will be submitted to an isokinetic muscular evaluation of the trunk extensor and flexor muscles and knee extensors and flexor performed in a Cybex Norm isokinetic dynamometer (Cybex Inc., Ronkonkoma, NY, USA).
Parkinson's Disease Questionnaire (PDQ-39) | 3 months
  The PDQ-39 will be applied to assess the patient's perception of quality of life, participation and restrictions resulting from the disease. The PDQ-39 is the most used disease-specific quality of life assessment tool in PD. The questionnaire consists of 39 questions covering the themes: mobility, activities of daily living, emotional well-being, social support, bodily discomfort, stigma, cognition and communication. The individual identifies how often in the last month he found himself in the situations mentioned. The options are never (0 points), rarely (1 point), sometimes (2 points), often (3 points), and always (4 points). Between 0 and 100, the lowest score corresponds to the highest quality of life.
Sit-and-Reach test | 3 months
  Muscle flexibility will be assessed by the Sit-and-Reach (SR) test, in which the patient, sitting with legs extended and feet resting on a box, leans forward keeping arms extended and knees straight. The greatest distance reached will be recorded in centimeters (cm).
30-second sit-to-stand test | 3 months
  The 30-second sit-to-stand test (STS) assesses functional capacity by recording the number of repetitions completed within a set time. Participants will begin by sitting in a 17-inch-high chair with their arms crossed in front of their chest and perform the sit-to-stand cycles as quickly as possible. They will be instructed to stand fully upright and to touch the seat each time they sit down again.

SECONDARY OUTCOMES:
Thigh and quadriceps muscle quality by specific tension and echo intensity | 3 months
  Muscle quality will be assessed using three distinct specific methods. First, quadriceps specific tension (QST) will be calculated as knee extension PT (N.m) divided by the sum of RF, VI, and VL MT (mm). Second, thigh specific tension will be calculated by the sum of knee flexion and extension PT (N.m) divided by TFFM (kg), assessed by DXA. Third and last, Echo Intensity (EI) will be calculated as the mean pixel value ranging from 0 (black) to 255 (white).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No